CLINICAL TRIAL: NCT05661916
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Subcutaneously Administered ALN-TTRSC04 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ALN-TTRSC04 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-TTRSC04-001
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin-Mediated Amyloidosis
Keywords: ATTR amyloidosis; siRNA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALN-TTRSC04 (Experimental): Participants will be administered a single dose of ALN-TTRSC04.
  Interventions: Drug: ALN-TTRSC04
- Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-TTRSC04 — ALN-TTRSC04 will be administered by subcutaneous (SC) injection.
  Arms: ALN-TTRSC04
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of single ascending doses of ALN-TTRSC04.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.0 kg/m^2 and ≤30 kg/m^2 assessed at Screening.

Exclusion Criteria:

* Has an estimated glomerular filtration rate (eGFR) <90 mL/min/1.73m^2 at screening.
* Has alanine aminotransferase (ALT), aspartate aminotransferase (AST) or direct bilirubin above the upper limit of normal (ULN).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | Up to 20 months

SECONDARY OUTCOMES:
Change from Baseline in Serum Transthyretin (TTR) Levels Over Time | Up to 18 months
Maximum Observed Plasma Concentration (Cmax) of ALN-TTRSC04 | Day 1 up to Day 4
Time to Maximum Observed Plasma Concentration (Tmax) of ALN-TTRSC04 | Day 1 up to Day 4
Area Under the Concentration-time Curve (AUC) of ALN-TTRSC04 | Day 1 up to Day 4
Fraction of ALN-TTRSC04 Excreted in the Urine (fe) | Up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (1):
- Clinical Trial Site, London, LND, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232